CLINICAL TRIAL: NCT02523690
Title: Evaluating Lorcaserin Drug Therapy For ICU-Acquired Weakness: A Pilot Randomized Trial
Brief Title: Evaluating Muscle Weakness Improvement With Lorcaserin in ICU
Acronym: EMILI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment of eligible patients
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00072940; UL1TR001079 (NIH)
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Muscle Weakness; Sepsis
MeSH Terms: conditions — Muscle Weakness; Sepsis | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Lorcaserin will be administered as a single dose on day 1 and day 3 to participants in this arm.
  Interventions: Drug: Lorcaserin
- Control (Placebo Comparator): Placebo will be administered as a single dose on day 1 and day 3 to participants in this arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorcaserin — 10 mg, oral or enteral, single dose. 30 mg, oral or enteral, single dose two days later
  Arms: Intervention
Drug: Placebo — Oral or enteral, single dose. Oral or enteral, single dose two days later
  Arms: Control

SUMMARY:
ICU acquired muscle weakness is a significant problem in patients recovering from critical illness. This trial will evaluate the safety and efficacy of a drug in improving muscle weakness in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Sepsis [ ≥2 Systemic Inflammatory Response Syndrome (SIRS) Criteria AND known or suspected infection]
* Muscle weakness [Medical Research Council sum score <48/60 or handgrip strength <11 kg in men and <7 kg in women]
* Obey Commands [Score for DeJonghe Awakening Score of ≥3/5]

Exclusion Criteria:

* Severe renal insufficiency [Creatinine Clearance <30 mL/min - or receiving dialysis]
* Acute infectious or auto-immune hepatitis, acute liver failure or a history of cirrhosis without liver transplant
* History of psychosis
* Bradycardia, or 2nd or 3rd degree Atrio-Ventricular block without pacemaker
* History of valvular heart disease without valve replacement
* History of priapism
* Pre-existing cognitive impairment
* Receiving drugs with serotonergic effects and/or CYP2D6 substrates which cannot be substituted stopped or titrated.
* Receiving Sulfonylurea medication at the time of the study
* Prior neuromuscular or central nervous system disease, including pre-existing neuropathy
* Inability to perform study's muscle strength assessments based on patient's baseline status prior to hospital admission
* Unable to receive, or unlikely to absorb study drug (e.g. bowel obstruction, ischemia, or infarction; short gut syndrome)
* Body mass index >40
* Patient not expected to survive >4 days
* Pregnancy or lactation
* Allergy to lorcaserin or lorcaserin taken in the prior 7 days
* Enrolled in another interventional drug or physical rehabilitation trial
* Physician declines for patient to be enrolled
* Patient or proxy declines consent
* Unable to reach proxy for consent
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale M Needham, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (19.8) | 56.0 (18.4) | 60.6 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Handgrip Strength as Measured by Hand Dynamometer
Description: Hand grip strength measured using a dynamometer (measured in kilograms, then compared to age- and sex-matched population norms to yield percent predicted strength - higher is better)
Time Frame: Baseline and 2 to 6 hours after administration of 30mg lorcaserin/placebo
Measure: Mean (Standard Deviation); unit: percent of predicted strength
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
percent of predicted strength | 0.67 (2.93) | 1.75 (1.06)

2. Secondary Outcome: Change in Handgrip Strength as Measured by Hand Dynamometer
Description: as for outcome 1
Time Frame: Baseline and 2 to 6 hours after administration of 10mg lorcaserin/placebo
Measure: Mean (Standard Deviation); unit: percent of predicted strength
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
percent of predicted strength | -3.83 (1.89) | 2.25 (0.35)

3. Secondary Outcome: Change in Manual Muscle Strength as Measured by the Medical Research Council (MRC) Score
Description: Measuring strength of 6 muscle groups in arms and legs using Medical Research Council composite score (each muscle group scored from scale of 0 [no visible or noticeable contraction] to 5 [maximum strength] and the sum of the scores for the 6 muscle groups equate to a composite score ranging from 0 to 60, higher score is better).
Time Frame: Baseline and 2 to 6 hours after administration of 30mg lorcaserin/placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
score on a scale | 0.33 (3.5) | 3.50 (2.12)

4. Secondary Outcome: Change in Manual Muscle Strength as Measured by the Medical Research Council (MRC) Score
Description: as for outcome 3
Time Frame: Baseline and 2 to 6 hours after administration of 10mg lorcaserin/placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
score on a scale | 1.00 (1.73) | 0.50 (0.71)

5. Secondary Outcome: Change in Quadriceps Strength as Measured by Handheld Dynamometer
Description: Strength (in kilograms) - measured via handheld dynamometry of quadriceps muscle.
Time Frame: Baseline and 2 to 6 hours after administration of 30mg lorcaserin/placebo
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
kilograms | -0.23 (1.83) | 4.15 (2.19)

6. Secondary Outcome: Change in Quadriceps Strength as Measured by Handheld Dynamometer
Description: Strength (in kilograms) - measured via handheld dynamometry of quadriceps muscle.
Time Frame: Baseline and 2 to 6 hours after administration of 10mg lorcaserin/placebo
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3 | 2
kilograms | 0.02 (1.23) | 2.13 (5.76)

ADVERSE EVENTS:
Time Frame: While admitted in hospital. For the 5 participants in this study, the mean number of days between enrollment and hospital discharge is 17.6 days (standard deviation 12.9 days)
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT02523690/Prot_SAP_000.pdf